CLINICAL TRIAL: NCT00295399
Title: Telerehabilitation for the Hand and Arm After Stroke and Traumatic Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ono Academic College (Other)
Responsible Party: Dr. Heidi Sugarman, Principal Investigator, Ono Academic College
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JTRS001
Record Dates: First submitted 2006-02-21; First posted 2006-02-23 (Estimated); Last update posted 2008-08-13 (Estimated); Status verified 2008-08

CONDITIONS: Cerebrovascular Accident; Traumatic Brain Injury
Keywords: cerebrovascular accident; traumatic brain injury; stroke; telerehabilitation
MeSH Terms: conditions — Stroke; Brain Injuries, Traumatic

INTERVENTIONS:
Device: The Jerusalem Telerehabilitation System

SUMMARY:
The goal of this project is to develop a low-cost, user-friendly, portable telerehabilitation system for physical therapy of the upper limb after stroke or traumatic brain injury. The system is based on the use of a commercially available force feedback joystick and will work with an ordinary home PC and a standard high-speed internet connection. Using the joystick, the patient will perform exercises designed to aid in recovering motor function of the hand and arm. The joystick will be programmed to either assist or resist the patient's movements. The system will include sophisticated analysis of patient status and progress to provide the therapist and physician with detailed information. In the first phase of the study, we will develop the system in cooperation with the physical therapy staff and other rehabilitation specialists. The investigators will examine the usability, comfort, safety and therapeutic benefit of the system. In the second phase of the study, the investigators will employ the system in patients' homes, using the internet to connect to rehabilitation specialists in the clinic. The study hypothesis is that it is possible to adapt commercially available, low cost gaming equipment such as force feedback joysticks to provide therapy for patients in their own homes, and that patients will be able to work with this system and will find it enjoyable and helpful for recovering motor function.

ELIGIBILITY:
Inclusion Criteria:

* Post-cerebrovascular accident or post-traumatic brain injury
* In medically stable condition
* Resident in Israel

Note: In addition there will be healthy, age-matched volunteers

Exclusion Criteria:

* History of psychiatric illness
* Grade of less than 23 in the Mini-Mental Test
* Inability to understand informed consent form
* Inability to follow 3-step instructions
* Pregnancy
* Receptive aphasia

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Modified motor assessment scale
Kinematic analysis
Feedback questionnaires for patients, therapists and caretakers

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Sugarman, Ph.D., Study Chair — Ono Academic College; Joseph Tiran, PhD, Principal Investigator — Ben Gurion University, Beer Sheva, Israel; Ehud Dayan, BSc, Principal Investigator — Sonarion Hadassah Virtual Reality Center
Locations (2):
- Israel (2):
  - Hadassah Medical Organization, Jerusalem
  - Chaim Sheba Medical Center, Tel Litwinsky

REFERENCES:
- [Background] Sugarman H, Dayan E, Weisel-Eichler A, Tiran J. The Jerusalem TeleRehabilitation System, a new low-cost, haptic rehabilitation approach. Cyberpsychol Behav. 2006 Apr;9(2):178-82. doi: 10.1089/cpb.2006.9.178. PMID 16640475